CLINICAL TRIAL: NCT02063282
Title: The Risk for Clostridium Difficile Colitis During Hospitalization in Asymptomatic Carriers
Status: Completed | Type: Observational
Sponsor: Amos Yinnon (Other)
Responsible Party: Sponsor-Investigator, Amos Yinnon, Professor, Shaare Zedek Medical Center
Organization: Shaare Zedek Medical Center (Other)
Other Study IDs: ShaareZMC
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Clostridium Difficile; Colitis
Keywords: Asymptomatic; Carriage; Colonization; Clostridium difficile; Colitis; Rectal swab
MeSH Terms: conditions — Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Clostridium difficile carriers
- Clostridium difficile non carriers

SUMMARY:
The investigators hypothesize that development of symptoms characteristic of Clostridium difficile infection will be 2-3 times higher in asymptomatic carriers, compared to that of non carriers and expect to find risk factors for development of symptomatic clostridium difficile.

ELIGIBILITY:
Inclusion Criteria:

* History of hospitalization in recent year, residence of a nursing home or institutions
* Expected more than 48 hours hospitalization

Exclusion Criteria:

* Colitis/ diarrhea
* Rectal swab performed ≥48 hrs post arrival to hospital.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Newly admitted patients in the Emergency Department and Internal wards, .
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Development of colitis | Daily follow-up
  participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
  Patients' file will be reviewed and the next signs and symptoms will be recorded: abdominal pain, diarrhea, fever and leukocytosis.

SECONDARY OUTCOMES:
Duration until development of colitis | Daily follow-up
  participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
  Patients' file will be reviewed and the next signs and symptoms will be recorded: abdominal pain, diarrhea, fever and leukocytosis.
Severity of colitis | Daily follow-up
  participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
  Patients' file will be reviewed and the next signs and symptoms will be recorded: abdominal pain, diarrhea, fever and leukocytosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No